CLINICAL TRIAL: NCT06882759
Title: Relationship of Point-of-care Coagulation Assays with Clinical Outcomes in Cardiac Surgery: a Retrospective Cohort Study
Status: Not yet recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 24-5983
Record Dates: First submitted 2025-03-10; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Cardiac Surgery Requiring Cardiopulmonary Bypass
Keywords: cardiac surgery; viscoelastic testing; point-of-care; ROTEM; cardiopulmonary bypass; bleeding
MeSH Terms: conditions — Hemorrhage | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cardiac surgery patients: Adult patients undergoing cardiac surgery on cardiopulmonary bypass at Toronto General Hospital
  Interventions: Other: No intervention (observational study)

INTERVENTIONS:
Other: No intervention (observational study) — This is an observational study. No intervention.

SUMMARY:
The goal of this observational study is to determine the relationship of ROTEM point-of-care coagulation assay parameters with excessive bleeding and clinical outcomes in patients undergoing cardiac surgery at Toronto General Hospital. The main questions it aims to answer are: i) How well does viscoelastic testing (VET) predict the clinical outcome of excessive bleeding in cardiac surgery? ii) Which VET parameters have the greatest accuracy for identification of patients who will have excessive bleeding? iii) 3) What is the prognostic value of abnormal VET parameters with other clinical outcomes after cardiac surgery?

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years old
* Underwent a cardiac surgical procedure with cardiopulmonary bypass

Exclusion Criteria:

- Did not undergo viscoelastic testing during surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac surgery with cardiopulmonary bypass at Toronto General Hospital
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Excessive bleeding | From the end of bypass to the end of postoperative day-1 (POD1)
  Measured by the universal definition of perioperative bleeding (UDPB) scale

SECONDARY OUTCOMES:
Transfusion rate | 1) From time of entry to operating room (OR) to the end of post-operative day-1 (POD1) and post-operative day-7(POD7). 2) from end of cardiopulmonary bypass (CPB) to the end of post-operative day-1 (POD1) and post-operative day-7 (POD7)
  Incidence and amount of transfusion of allogeneic blood products and factor concentrates

CONTACTS AND LOCATIONS:
Overall Officials: Keyvan Karkouti, Principal Investigator — University Health Network, Toronto

IPD SHARING:
Plan to Share IPD: No